CLINICAL TRIAL: NCT05940363
Title: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease With a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies Based on Multi-center Collaboration in China
Brief Title: The National Program for the Improvement of Management of Fetal Congenital Heart Disease in China
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yihua He,MD, Director of the Center for Maternal-Fetal Medicine of Fetal Heart Disease, Beijing Anzhen Hospital
Other Study IDs: MCCDTP-CHD
Record Dates: First submitted 2023-07-02; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Congenital Heart Disease in Pregnancy; Prenatal Diagnosis; Fetal Echocardiography
Keywords: Congenital Heart Disease; Prenatal diagnosis; Fetal Echocardiography; Maternal-fetal medicine; Digital health technologies
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Liaoning Provincial Maternal and Child Health Hospital: Liaoning Provincial Maternal and Child Health Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Shenyang Maternal and Infant Hospital: Shenyang Maternal and Infant Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Guangdong Women and Children's Hospital: Guangdong Women and Children's Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Guangzhou Women and Children's Medical Center: Guangzhou Women and Children's Medical Center
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Guangdong Provincial People's Hospital: Guangdong Provincial People's Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Shandong Maternal and Child Health Hospital: Shandong Maternal and Child Health Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Fujian Provincial Maternal and Child Health Hospital: Fujian Provincial Maternal and Child Health Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Maternal and Child Health Hospital of Hubei Province: Maternal and Child Health Hospital of Hubei Province
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Anhui Provincial Maternal and Child Health Hospital: Anhui Provincial Maternal and Child Health Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Peking University First Hospital, Ningxia Women and Children's Hospital: Peking University First Hospital, Ningxia Women and Children's Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies
- Sichuan Maternal and Child Health Hospital: Sichuan Maternal and Child Health Hospital
  Interventions: Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies

INTERVENTIONS:
Combination Product: Improvement on Prenatal Screening and Treatment Capabilities for Congenital Heart Disease with a Comprehensive Diagnosis and Treatment Program Incorporating New Technologies — To investigate and evaluate the capacity of prenatal screening, diagnosis and counseling for fetal heart disease based on medical institutions; Improving capacity for prenatal screening, diagnosis and counselling through integrated products embedded with new technologies.

SUMMARY:
To investigate and evaluate the capacity of prenatal screening, diagnosis and counseling of congenital heart disease in medical institutions in China, in order to understand the current status and existing problems of prenatal prevention and treatment capacity of congenital heart disease in China, and to obtain corresponding baseline data, so as to provide scientific basis for further improving prenatal screening and diagnosis policies in China.

DETAILED DESCRIPTION:
With the rapid development of medical imaging technology, the role of ultrasound screening and diagnosis in the prevention and treatment of birth defects is increasingly prominent. Early screening, classified diagnosis, and standardized consultation are the basis for effective prevention and treatment of congenital heart disease. Due to the uneven development of medical resources and medical service levels in the eastern, central, and western regions of China, as well as between urban and rural areas, the ability of prenatal ultrasound screening, diagnosis, and clinical consultation varies greatly, and there is a lack of relevant clinical research data, which makes it difficult to adopt effective intervention measures. This study aims to investigate and analyze the prenatal screening, diagnosis, and consultation abilities of medical personnel in different regions, evaluate the current status and problems of congenital heart disease abilities in various regions, explore a multidisciplinary transfer consultation integrated service mechanism, strengthen comprehensive prevention and control abilities, ensure maternal and infant health.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women and fetuses who underwent prenatal ultrasound examination in the above hospitals were enrolled

Exclusion Criteria:

* Pregnant women not willing to cooperate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women and physicians performing prenatal screening and diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The integrity rate of the multi-view acquisition | From June 2023 to Oct 2023
  The integrity rate of the multi-view acquisition
Negative coincidence rate congenital heart disease screening | From June 2023 to Oct 2023
  Negative coincidence rate congenital heart disease screening
Positive coincidence rate of congenital heart disease screening | From June 2023 to Oct 2023
  Positive coincidence rate of congenital heart disease screening
The coincidence rate of multidisciplinary consultation | From June 2023 to Oct 2023
  The coincidence rate of multidisciplinary consultation

CONTACTS AND LOCATIONS:
Overall Officials: Yihua He, MD, Study Chair — Beijing Anzhen Hospital

IPD SHARING:
Plan to Share IPD: Undecided